CLINICAL TRIAL: NCT05498961
Title: The Effect of Gallstone Characteristics for the Severity of Acute Gallstone Pancreatitis
Brief Title: The Effect of Gallstone Characteristics for the Severity of Gallstone Pancreatitis
Status: Completed | Type: Observational
Sponsor: Hepatopancreatobiliary Surgery Institute of Gansu Province (Other)
Responsible Party: Principal Investigator, Wenbo Meng, Professor of surgery, Hepatopancreatobiliary Surgery Institute of Gansu Province
Other Study IDs: acute gallstone pancreatitis
Record Dates: First submitted 2022-08-10; First posted 2022-08-12 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Acute Gallstone Pancreatitis
Keywords: Pancreatitis; Gallstone; Severity
MeSH Terms: conditions — Pancreatitis; Gallstones

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Gallstone characteristics — stone size, number, the thickness

SUMMARY:
The purpose of this study was to determine the effect of gallstone characteristics for the severity of acute gallstone pancreatitis (GSP)

DETAILED DESCRIPTION:
The timing of cholecystectomy is closely related to the severity of acute gallstone pancreatitis (GSP). The effect of gallstone characteristics (including stone size, number, etc.) for the severity of GSP are currently unknown.

ELIGIBILITY:
Inclusion Criteria:

* Acute gallstone pancreatitis (GSP) patients.

Exclusion Criteria:

* Pancreatitis with bile duct stones, trauma, drugs, and surgery;
* Recurrent gallstone pancreatitis;
* Combined with other malignant tumors, such as liver cancer, cholangiocarcinoma, pancreatic cancer, gastric cancer, Hematologic tumor, and lymphoma;
* Previous hepatobiliary and pancreatic surgery, Organ transplantation;
* Intestinal obstruction or other obstructive diseases;
* Chronic pancreatitis or pancreatic duct stones;
* Thrombotic disease;
* Alcoholic pancreatitis and hyperlipidemia pancreatitis.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute gallstone pancreatitis patients
Sampling Method: Probability Sample
Enrollment: 301 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2023-09-24 (Actual); Study Completion 2023-09-24 (Actual)

PRIMARY OUTCOMES:
Number of severity of GSP patients | 1 month
  Based on the 2012 Atlanta International Consensus, Mild acute pancreatitis (MAP) is defined as no organ failure and no local or systemic complications. Moderate to severe acute pancreatitis (MSAP) refers to patients with organ failure, local complications, or aggravated complications. Severe acute pancreatitis (SAP) is defined as persistent organ failure for more than 48 hours.

SECONDARY OUTCOMES:
Modified computed tomography severity index (MCTSI) score | 1 month
  Without knowing the prognosis, two radiologists with eight and ten years of experience independently scored the severity of GSP through the MCTSI score and reached an agreement through discussion when there was disagreement.
Gallstone size | 1 month
  The diameter of the stones
Number of stones | 1 month
  The number of gallstones

CONTACTS AND LOCATIONS:
Overall Officials: Wenbo Meng, M.D.,Ph.D, Principal Investigator — LanZhou University
Locations (1):
- Hepatopancreatobiliary Surgery Institute of Gansu Province, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: No
If patients permitted

REFERENCES:
- [Background] Yadav D, Lowenfels AB. The epidemiology of pancreatitis and pancreatic cancer. Gastroenterology. 2013 Jun;144(6):1252-61. doi: 10.1053/j.gastro.2013.01.068. PMID 23622135
- [Background] Boxhoorn L, Voermans RP, Bouwense SA, Bruno MJ, Verdonk RC, Boermeester MA, van Santvoort HC, Besselink MG. Acute pancreatitis. Lancet. 2020 Sep 5;396(10252):726-734. doi: 10.1016/S0140-6736(20)31310-6. PMID 32891214
- [Derived] Ma Y, Yue P, Zhang J, Yuan J, Liu Z, Chen Z, Zhang H, Zhang C, Zhang Y, Dong C, Lin Y, Liu Y, Li S, Meng W. Early prediction of acute gallstone pancreatitis severity: a novel machine learning model based on CT features and open access online prediction platform. Ann Med. 2024 Dec;56(1):2357354. doi: 10.1080/07853890.2024.2357354. Epub 2024 May 30. PMID 38813815